CLINICAL TRIAL: NCT06965725
Title: Evaluation of a Novel Paired-Ring Mitral Annuloplasty Sizing Method and Device
Brief Title: Paired-Ring Mitral Annuloplasty Ring Sizing Device
Status: Active, not recruiting | Type: Observational
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Nikola Dobrilovic, MD, Endeavor Health
Other Study IDs: EH23-243
Record Dates: First submitted 2025-04-24; First posted 2025-05-11 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-05

CONDITIONS: Heart Valve Diseases
Keywords: Annuloplasty Ring; Sizing methods
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Annuloplasty ring sizing tool: A single time use of a novel sizing tool for mitral valve repair surgery
  Interventions: Device: Annuloplasy ring sizing device

INTERVENTIONS:
Device: Annuloplasy ring sizing device — A single time use of a novel sizing tool for mitral valve repair surgery (used ONLY in an observational capacity - this device does NOT influence decision-making during the conduct of the operation in any way).

SUMMARY:
The purpose of this study is to evaluate a novel paired-ring mitral annuloplasty sizing system in humans.

DETAILED DESCRIPTION:
This is a pilot feasibility study of an investigational device. The proposed device is designed to be used as a temporary, disposable tool that will guide final ring size selection during mitral valve repair surgery. This device enables the direct measurement of the mitral valve opening. Currently, sizing tools for mitral annuloplasty ring implantation has provide only a rough estimate. The field of cardiac surgery is in need of a precise technique to accomplish the important task of correctly selecting an annuloplasty ring for implantation.

ELIGIBILITY:
Inclusion Criteria:

1. All patients scheduled for mitral repair surgery
2. Age 18 years or older

Exclusion Criteria:

1. Adults unable to consent,
2. Pregnant women and prisoners.
3. Emergency operations and those patients in whom mitral repair is not performed in a meaningful way, requiring mitral replacement instead, will be excluded.
4. Presence of acute endocarditis infection during the initial screening process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing mitral valve repair.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Mitral leaflet coaptation length. | During surgery, immediately prior to prosthesis implantation.
  Direct measurement of mitral leaflet coaptation length performed with the sizer in position, performed in mm using surgical (disposable) ruler.
Post-procedure, echocardiography measurements - mitral coaptation length. | After separation from cardiopulmonary bypass.
  Indirect measurement of mitral leaflet coaptation length (mm), using standard intraoperative trans-esophageal echocardiography (TEE) images (measurements performed postoperatively based on archived images).

CONTACTS AND LOCATIONS:
Overall Officials: Nikola Dobrilovic, MD, Principal Investigator — Endeavor Health
Locations (1):
- Endeavor Health, Glenview, Illinois, United States

IPD SHARING:
Plan to Share IPD: No